CLINICAL TRIAL: NCT03271905
Title: Influence of Mechanical Ventilation Modes on the Efficacy of Nebulized Bronchodilator in the Treatment of Patients With Obstructive Pulmonary Disease
Brief Title: Influence of Mechanical Ventilation Modes on the Efficacy of Nebulized Bronchodilator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Cibelle Andrade Lima, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CibelleAndrade
Record Dates: First submitted 2017-06-08; First posted 2017-09-05 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant is blind about the procedures. The investigator is blind about order of procedure and outcomes assessor is blind about procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pressure-controled-ventilation (PCV) (Experimental): Nebulization during mechanical ventilation on a pressure controled ventilation mode.
  Interventions: Drug: salbutamol sulfate and ipratropium bromide; Device: Mesh nebulization
- PCV and high PEEP (Experimental): Nebulization during mechanical ventilation on a pressure controled ventilation mode and PEEP = 15 cmH2O.
  Interventions: Drug: salbutamol sulfate and ipratropium bromide; Device: Mesh nebulization
- Pressure suport ventilation (PSV) (Experimental): Nebulization during mechanical ventilation on a pressure suport ventilation mode.
  Interventions: Drug: salbutamol sulfate and ipratropium bromide; Device: Mesh nebulization

INTERVENTIONS:
Drug: salbutamol sulfate and ipratropium bromide — Nebulization with salbutamol sulfate and ipratropium bromide during mechanical ventilation.
Device: Mesh nebulization — Nebulization with Mesh device.

SUMMARY:
Aerosol therapy is widely used in intensive care in critically ill patients that use mechanical ventilation (MV). However, there is a lack of standardization about aerosol performance in this group of patients. Thus, this study aims to evaluate the effect of nebulization performed in different ventilatory modes on lung function and regional pulmonary distribution of critical patients with chronic obstructive pulmonary disease. It is a clinical trial, crossover, randomized, controlled and blind. Three interventions with bronchodilators will be performed: in the Pressure Controlled Ventilation mode (PCV) with positive end expiratory pressure (PEEP) = 85% of autoPEEP, in the PCV mode with PEEP = 15 cmH2Oand in the Pressure Support Mode (PSV). Pulmonary function data will be evaluated through Electrical Impedance Tomography to evaluate the efficacy of the bronchodilator in different ventilatory modes.

DETAILED DESCRIPTION:
2. OBJECTIVES

2.1 Primary

• To evaluate the influence of mechanical ventilation modes in the efficacy of nebulized bronchodilator in ventilator dependent patients with obstructive pulmonary disease.

2.2 Secondary

* To compare regional ventilation distribution through Ventilation Surface Area (VSA) and Tidal Impedance Variation (TIV or ∆Z) by electrical impedance tomography (EIT) before, immediately after, after 1hour (h), 2h and 3h of nebulized bronchodilator in pressure controlled ventilation (PCV) with and without sedative drugs, and during pressure support ventilation (PSV).
* To compare the peak expiratory flow (PEF), change in End-Expiratory Lung Volume (dEELV), Respiratory Compliance (Crs) and Resistance (R), before, immediately after, after 1h, 2h and 3h of nebulized bronchodilator by monitoring airway pressure and EIT in ventilator modes PCV, with and without sedative drugs and PSV .
* To compare the ventilator modes on the VSA, ∆Z, PEF, dEELV and Crs after nebulized bronchodilator and the duration of its effects during mechanical ventilation.
* To compare two different level of PEEP during nebulized bronchodilator on PCV mode while the patient stay with sedative drugs.

  3. METHODS

3.1 Study design This is a randomized crossover, blinded clinical trial. The randomization procedure will be a simple randomization by random number table. In order to improve reliability, not transparent sealed envelopes for blind allocation will be used.

3.2 Local and study period This is a multicenter study that involve the following hospitals: Hospital Miguel Arraes - PE and Real Hospital Português de Beneficência em Pernambuco- PE. All hospitals are located in the metropolitan region of Recife, Pernambuco, Brazil and the study will be conducted from February 2016 to December 2019.

3.3 Sample The study population consist of patients with obstructive pulmonary disease admitted to intensive care unit for MV support who meet the inclusion criteria.

3.4 Sample size Patients will be identified by a daily telephone calls to the ICUs each morning for data collection. Potential candidate patients will be screened for inclusion and exclusinon criteria, after the identification of eligible patients. After consent is obtained, the research team goes to the ICU to start collecting data. The sample size will be calculated by statistical procedures after conducting a pilot study of 10 patients.

3.5 Technical procedures and tools for data collection

Prior to starting the intervention, clinical and demographic data will be collected according to the evaluation form, ( Appendix 2). After that, patients will be receive each of 4 interventions, with a minimum of 4 hours between bronchodilator administration to allow for washout.

3.5.1. Intervention Protocol 3.5.1.1. Step 1: Nebulization during Pressure Controlled Ventilation (PCV) Mode Initially the patient will be accessed when he still sedated. Two intervention will be done with a PCV mode in two different ways and the order of the procedures will be randomized.

One nebulization will be done with a standard PCV mode and parameters will be setted as follows: sufficient Δ pressure to maintain the patient's tidal volume (vt) at 6 / kg ideal weight, respiratory rate (RR) at 12 bpm, inspiratory time (Ti) up to 1 second, maintain Ti / Ttot 0.3 - 0.4 without causing dynamic AutoPEEP, decreasing waveform flow and PEEP level of 85% from static autoPEEP.

Other nebulization will be done also in PCV mode with same parameters, but the level of PEEP will be increased to 15 cmH2O. Between this two interventions will be given 4 hours for washout.

After this, we will talk to the medical staff to interrupt sedation, will be given 3 hour for wash out to start de Step 2.

3.5.1.2. Step 2: Nebulization During Pressure Support Ventilation (PSV) With a clinical progression of the patient, a 4th evaluation will be done on the first day when the patient achieve PSV mode. In this ventilation mode the patient will control the Ti, Ttot, RR and inspiratory flow so it will be set only one Δ pressure for the patient to support a Vt of 6 ml/kg. The lowest minimum value of Δ P is 10 cmH2O and the end of inspiratory phase will be determined by a decrease at 25% of the patient peak inspiratory flow.

3.5.2 Nebulization Protocol

Nebulized bronchodilator drugs will be Salbutamol Sulfate (aerolin nebulis) and ipratropium bromide (atrovent) diluted in a saline solution (saline 0.9%) in 3 ml. The vibrating Mesh nebulizer (Aeroneb Pro-X, Galway, Ireland) will be placed in the inspiratory circuit of the MV immediately before 'Y' piece using a 22 mm T adapter. The nebulizer is operated by an electric controller connected mains power. The vibrating Mesh produces aerosol with an average particle size of 5 μm and will remain on continuously until the end of nebulization.

If a heat moisture exchanger (HME) is used during mechanical ventilation, it must be removed from between the nebulizer and airway before nebulization so that it does not filter out and reduce aerosol delivered.

3.5.3 Evaluation by Electrical Impedance Tomography. TIE is a tool of obtaining transverse plane image of any section of the human body by means of low-power electric current. The image is obtained from the electric current or potential detected on the surface of the evaluated area, where each "pixel" image is its impedance or resistivity. Thus, when used in thoracic follow-up, the EIT is able to evaluate the aeration and ventilation of the patient through the following variables: distribution of regional lung ventilation by Tidal Impedance Variation (ΔZ), Ventilation Surface Area (VSA), Percentage of Recruitable Lung (PRLV), Change in End-Expiratory Lung Volume (dEELV) and Respiratory Compliance (Crs) .

Initially, to evaluate the acute pulmonary impact of nebulizer bronchodilator on different ventilatory modes, EIT will be be performed before and immediately after the aerosol administration and repeated with each ventilation mode. Furthermore, the duration of nebulization effect will be evaluated by performing EIT after 1, 2 and 3h in each ventilation mode. There will be a > 4 hour washout between bronchodilator administrations.

An impedance tomography (ENLIGHTER, Timpel, Brazil) will be used with the patient in supine position with a bed elevation of 45◦, so a belt with 32 electrodes will be applied to the chest, in the position corresponding to the 4th - 5th intercostal space on a shaved skin. Electrodes have to be positioned for reading electrocardiograms and a flow sensor that should be attached to the endotracheal tube. After this procedures recording data starts for 3 minutes.

For image acquisition, harmless electrical currents (5-8 nA, 125 KHz) will be injectates through electrode pairs in rotating sequence, and the potential differences Will be captured in other non injetantes electrode. Variations in thoracic impedance will be evaluated through a LabView software (National Instruments, USA) and the data is recorded in separate files for patients for further analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients with asthma or chronic obstructive pulmonary disease (COPD) Invasive mechanical ventilation Hemodynamically stable

Exclusion Criteria:

Prescribed metered dose inhaler (MDI) or intravenous bronchodilators Undrained pneumothorax Bronchopleural fistula Chest trauma Tracheoesophageal fistula Tracheal granulomas Tracheal stenosis PEEP dependence

Contraindicated disconnection of the MV

Endotracheal tube diameter less than 7.5

Do not make part of the protocol of daily sedation

No regular ventilatory drive when with out sedation

Do not reach a minimum tidal volume 6 ml/kg with a maximum peak pressure (PIP) of 35 cmH2O (centimeter of water) during MV.

Do not use the same MV modes that will be tested in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in tidal Impedance Variation | change from baseline immediately after and at 1, 2, 3 hour of nebulized bronchodilator
  compare regional ventilation distribution by electrical impedance tomography

SECONDARY OUTCOMES:
Change in compliance of respiratory sistem (cmH2O) | change from baseline immediately after and at 1, 2, 3 hour of nebulized bronchodilator
  Compare results evaluated by lung mechanics evaluation
Change in peak expiratory flow (lpm) | change from baseline immediately after and at 1, 2, 3 hour of nebulized bronchodilator
  Compare results evaluated by EIT
Change in End-Expiratory Lung Volume | change from baseline immediately after and at 1, 2, 3 hour of nebulized bronchodilator
  Compare results evaluated by EIT

CONTACTS AND LOCATIONS:
Locations (1):
- Cibelle Andrade Lima, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No